CLINICAL TRIAL: NCT06676228
Title: Fear of Cancer Recurrence Therapy (FORT): Turkish Cultural Adaptation and Implementation Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Psiko-Onkologlar Dernegi (Turkish Psycho-Oncological Association) (Unknown); Oz Psikolojik Danismanlik Merkezi (Oz Psychological Consultancy) (Unknown)
Responsible Party: Principal Investigator, ASLI EYRENCI, Assist. Prof., Maltepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023/15-11
Record Dates: First submitted 2024-10-30; First posted 2024-11-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Self Efficacy; Anxiety; Depression Not Otherwise Specified; Fear of Cancer Recurrence; Cancer Coping; Quality of Life (QOL); Intolerance of Uncertainty
Keywords: FORT; Fear of cancer recurrence; Turkish; Fear of cancer recurrence therapy; breast cancer; cancer survivor
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms | interventions — Cognitive Behavioral Therapy; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Group leaders/care providers and investigators know the group assignments but the participants do not know which group they were assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): FORT consists of 6 sessions in total, the scopes of the sessions are detailed below:
  Session 1 (Acquiring new skills to cope with Fear of Cancer Recurrence (FCR)) HOMEWORK: Daily practice of progressive muscle relaxation exercise; creation of a thought record
  Session 2 (Providing information on symptoms of cancer recurrence and increasing tolerance to uncertainty) HOMEWORK: Listening to recordings of relaxation exercises every day; practising self-calming, keeping a record of thoughts
  Session 3 (Developing coping skills) HOMEWORK: Practise guided imagery daily; debunk erroneous beliefs about the benefits of worrying; keep a thought log
  Session 4 (Deepening the underlying fears) HOMEWORK: Reading the worst case fear scenario every day, practising daily self-care and mindfulness practices
  Session 5 (Moving beyond specific fears) HOMEWORK: Writing goals and priorities for the future
  Session 6 (Review and conclusion) Reviewing all the discussed content
  Interventions: Behavioral: Fear of cancer recurrence therapy (FORT)
- Control Group (active comparator) (Active Comparator): The cognitive-behavioural therapy (CBT) oriented control group consisted of a total of 6 sessions. The scopes of the sessions are given in detail below.
  Session 1: Introduction and cancer-focused psychoeducation with CBT HOMEWORK: Keeping a thought diary
  Session 2: Addressing the underlying causes of thoughts HOMEWORK: Keeping a thought diary about underlying beliefs
  Session 3: Recognising conflicts HOMEWORK: Task: Keep a diary of thoughts about disagreements (what gives us pleasure and what we should master)
  Session 4: Effective communication techniques HOMEWORK: Keeping a diary about the use of the word "good enough"
  Session 5: Discussion of the definitions of anxiety and depression
  Session 6: Anger Management HOMEWORK: HOMEWORK: Keeping a diary about the use of the breathing exercise
  Interventions: Behavioral: cognitive-behavioural therapy (CBT) group

INTERVENTIONS:
Behavioral: Fear of cancer recurrence therapy (FORT) — FORT consists of 6 sessions in total, the scopes of the sessions are detailed below:
  Session 1 (Acquiring new skills to cope with Fear of Cancer Recurrence (FCR)) HOMEWORK: Daily practice of progressive muscle relaxation exercise; creation of a thought record
  Session 2 (Providing information on symptoms of cancer recurrence and increasing tolerance to uncertainty) HOMEWORK: Listening to recordings of relaxation exercises every day; practising self-calming, keeping a record of thoughts
  Session 3 (Developing coping skills) HOMEWORK: Practise guided imagery daily; debunk erroneous beliefs about the benefits of worrying; keep a thought log
  Session 4 (Deepening the underlying fears) HOMEWORK: Reading the worst case fear scenario every day, practising daily self-care and mindfulness practices
  Session 5 (Moving beyond specific fears) HOMEWORK: Writing goals and priorities for the future
  Session 6 (Review and conclusion) Reviewing all the discussed content
  Arms: Experimental Group
Behavioral: cognitive-behavioural therapy (CBT) group — The cognitive-behavioural therapy (CBT) oriented control group consisted of a total of 6 sessions. The scopes of the sessions are given in detail below.
  Session 1: Introduction and cancer-focused psychoeducation with CBT HOMEWORK: Keeping a thought diary
  Session 2: Addressing the underlying causes of thoughts HOMEWORK: Keeping a thought diary about underlying beliefs
  Session 3: Recognising conflicts HOMEWORK: Task: Keep a diary of thoughts about disagreements (what gives us pleasure and what we should master)
  Session 4: Effective communication techniques HOMEWORK: Keeping a diary about the use of the word "good enough"
  Session 5: Discussion of the definitions of anxiety and depression
  Session 6: Anger Management HOMEWORK: HOMEWORK: Keeping a diary about the use of the breathing exercise
  Arms: Control Group (active comparator)

SUMMARY:
This research consists of two phases. The aim of the first study is to adapt the group work module of Fear of Cancer Recurrence (FCR) for FCR in survivors of breast and ovarian cancer patients to the Turkish culture. For cultural adaptation, a process consisting of four stages is planned to be followed based on the World Health Organisation (WHO) and ecological validity model: 1) literature review; 2) translation of the intervention manual from English to Turkish and evaluation of the translation by experts; 3) cognitive interviews with ovarian and breast cancer patients and experts working in the field of psychooncology about the sections of the translated manual; and 4) an adaptation workshop where data from the previous stages were collected and analysed. The aim of the second study, 6-week, 120-minute FCR (n= 68) or CBT intervention (n= 68) group sessions with participants from ovarian and breast cancer patients. They will be completing questionnaires at baseline (T0), post-treatment right after treatment ends (T1), 3 months (T2), and 6 months (T3) post-treatment. A generalized linear model will be used for the analysis of collected data, incorporating customized analyses such as ANCOVA for repeated measures and analysis of variance for repeated measures. The primary outcome will be compared to the Fear of Cancer Recurrence Inventory (FCRI) total score and group differences in secondary outcomes.

With this project, it is aimed to bring the group intervention module for FCR, which is a common problem in surviving cancer patients that will greatly contribute to the psycho-oncology practice in Turkiye. In addition, it is thought that this project is important both because there is no study on cancer survivors and FCR in this context and cultural adaptation studies are crucially limited in Turkey.

DETAILED DESCRIPTION:
First Phase: Cultural Adaptation Study

The aim of this study is to adapt the group work module for Fear of Cancer Recurrence (FCR) in breast and ovarian cancer survivors to the culture of Turkey. In this direction, the following cultural adaptation steps will be followed, Theoretical background of the FCR:

1. Document Evaluation: In the first stage, a comprehensive literature review will be conducted to identify the interventions currently implemented in the field of mental health in Turkey for breast and ovarian cancer survivors.
2. Translation and Review: At this stage, the first translation and back-translation of the FCR patient handbook from English to Turkish will be carried out. It will also be evaluated in terms of ecological group modelling.
3. Cognitive Interviewing: In this phase, focus interviews will be conducted with experts and breast and ovarian cancer survivors to assess the comprehensibility, cultural and survivorship context of the NCT patient handbook.
4. Adaptation Workshop: In the final stage, a workshop will be held to evaluate the data obtained in the previous stages, make adaptations and suggested changes, and finalise the adapted protocol.

Second phase: Intervention Study

A randomised control group study will be conducted within Work Package 2. In the intervention group of the study, the adaptation of the FCR will be applied, and in the control group, Cognitive Behavioural Therapy (CBT) focused group application will be performed. This study is planned as a single-blind study (a study in which the group leaders know the group assignments but the group members do not know which group they are in).

Participants Participants are planned to consist of clients of Oz Psychological Consultancy Centre and people reached through cancer associations/patient groups. It is planned to give gift vouchers to the participants who will participate in the study. The decision to give gift vouchers was made in order to minimise potential drop-out rate in this project.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are under 18 years of age
* Participants whose primary treatment (chemotherapy, radiotherapy, surgery) has been completed (adjuvant treatment such as hormone therapy may be continued can be accepted into the study).
* Participants with stage I-III breast cancer and ovarian cancer who have completed treatment less than 5 years ago and whose disease is in remission.
* Participants who receive cut-off scores of 10 or above for the anxiety and 7 or above for the depression Hospital and Anxiety Scale.
* Participants who score 4 for depression and 5 for anxiety and distress for the Emotion Thermometer.

Exclusion Criteria:

* Participants over 65 years of age
* Participants who experience of recurrence/metastasis
* Participants who has mental retardation
* Participants who do not possess Turkish language skills
* Participants who have another comorbid physical illness that causes disability
* Participants who were diagnosed with a psychiatric disorder.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — People who were born with female genitals (vagina).
Enrollment: 100 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-26 (Actual); Study Completion 2025-09-26 (Actual)

PRIMARY OUTCOMES:
Decreased Fear of cancer recurrences scores | 3 months and 6 months
  Patients score will change for the Fear of Cancer Recurrence Inventory. There are seven sub-dimensions: triggers, violence, psychological distress, coping strategies, functional impairments, insight, and search for reassurance. The triggers sub-dimension contains eight items, the violence sub-dimension contains nine items, the psychological distress sub-dimension contains four items, the coping strategies sub-dimension contains nine items, the functional impairments sub-dimension contains six items, the insight sub-dimension contains three items, and the search for reassurance sub-dimension contains three items, totaling 42 items. Additionally, there are five sub-dimensions: triggers, functional impairments, higher-order cognitions related to relapse, emotion-focused coping strategies, and quality of life, consisting of 24 items evaluated using a four-point Likert scale. As the scores obtained from the scale increase, so does the Fear of Cancer Recurrence.

SECONDARY OUTCOMES:
Higher level of Cancer Coping | 3 months and 6 months
  Participants score will change at the cancer coping questionnaire (CCQ). There are 21 items within this scale. The scale assesses the personal dimension with scores ranging from 1 to 4. Higher scores on the scale indicate that the specified coping method is used more frequently.
Higher level of tolerance of uncertainty | 3 months and 6 months
  Participants score will change in Intolerance of Uncertainty Scale. This scale consists of 12 items measured by responses on a 5-point Likert scale, and it includes two sub-dimensions: "future anxiety" and "preventive anxiety." The total score that can be obtained from the scale ranges from 12 to 60. A high score on the scale indicates a high level of intolerance to uncertainty.
Higher level of Self Efficacy | 3 months and 6 months
  Participant score will change in Self-Efficacy for Managing Chronic Disease (SEMCD) scale. The scale consists of 6 items and is evaluated on a 10-point Likert scale, where "1" represents "not at all sure" and "10" represents "completely sure." As the score obtained from the scale increases, the individual's self-efficacy related to their chronic illness also increases.
Higher level of Quality of Life | 3 months and 6 months
  Participants score will change in EORTC QLQ-C30 - Quality of Life questionnaire. The scale consists of subscales that evaluate overall health status, functionality (including physical, role, emotional, cognitive, and social functioning), and the presence of symptoms, totaling 30 items. Low scores on the functional subscales indicate low quality of life, while low scores on the symptom subscale, which assesses symptoms such as fatigue, pain, nausea, and vomiting, indicate high quality of life. The first 28 items of the scale are evaluated using 4-point Likert response options, while the 29th and 30th items, related to overall health status, are assessed using 7-point Likert response options. The scores obtained from the scale range from 0 to 100 for each subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Asli Eyrenci, PhD, Principal Investigator — Istanbul Maltepe University; Ozan Bahcivan, PhD, Study Director — Turkish Psycho-Oncological Association (Psiko-Onkologlar Dernegi)
Locations (1):
- Istanbul Maltepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared for the following reasons:
  1. Sharing IPD can raise privacy issues among participants (patients), as it may contain sensitive personal information about participants that must be protected under ethical regulations.
  2. Participants may not have given consent for their data to be shared publicly or used beyond the initial study, leading to ethical concerns about data sharing.

REFERENCES:
- [Derived] Eyrenci A, Ertuna L, Bahcivan O. Preliminary Outcomes of a Culturally Adapted Fear of Recurrence Therapy (FORT) for Turkish Breast Cancer Survivors: A Randomized Controlled Trial. Psychooncology. 2025 Dec;34(12):e70345. doi: 10.1002/pon.70345. PMID 41318944